CLINICAL TRIAL: NCT06137586
Title: The Effect of Glucose-dependent Insulinotropic Polypeptide on the Alpha Cell Response to Hypoglycaemia in Patients with Type 1 Diabetes
Acronym: GIPHYPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, Principal investigator, MD, ph.d., University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GIPHYPO2022
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Type1diabetes; Hypoglycemia; Type 1 Diabetes
Keywords: Incretins; GIP; Glucose-dependent insulinotropic polypeptide; Alpha cell
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — gastric inhibitory polypeptide (1-30)

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, single-arm study. Each participant goes through five experimental days in a randomized order - acting as their own controls
Masking Description: The randomized order of infusions is blinded to both participant and investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infusion of GIP[1-42], GIP[1-30] or placebo (Experimental): This is a single arm study. All participants will go through all five experimental days in a randomized order. The interventions are A) 4pmol/kg/min GIP[1-42] B) 8pmol/kg/min GIP[1-42] C) 4pmol/kg/min GIP[1-30] D) 8pmol/kg/min GIP[1-30] E) Saline (placebo)
  Interventions: Other: Infusion of GIP[1-42], GIP[1-30] or placebo

INTERVENTIONS:
Other: Infusion of GIP[1-42], GIP[1-30] or placebo — This is a single arm study. All participants will go through all five experimental days in a randomized order. The interventions are A) 4pmol/kg/min GIP[1-42] B) 8pmol/kg/min GIP[1-42] C) 4pmol/kg/min GIP[1-30] D) 8pmol/kg/min GIP[1-30] E) Saline (placebo)

SUMMARY:
The goal of this clinical trial is to evaluate the effects of the hormone glucose-dependent insulinotropic polypeptide (GIP) and its two isoforms, GIP[1-30] and GIP[1-42], in patients with type 1 diabetes. The main question it aims to answer is:

• What dose and isoform of GIP can most potently stimulate glucagon secretion during low blood sugar in patients with type 1 diabetes?

Participants will go through 5 experimental days that are identical except for an intravenous infusion of either placebo (saline), high or low dose GIP[1-42] or high or low dose GIP[1-30]. On all days, blood sugar will be lowered to around 2.5mmol/l for around 20-30min.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, each participant giving written informed consent will participate in five double-blinded experimental days (Day A-E) in a randomized order. Each experimental day is identical except for an intravenous infusion of either placebo (saline), high (8pmol/kg/min) or low (4pmol/kg/min) dose GIP[1-42] or high (8pmol/kg/min) or low (4pmol/kg/min) dose GIP[1-30].

Each experimental day will consist of an induction period where the participant's blood sugar is adjusted to around 5-6mmol/l with either insulin or glucose. Then the infusion of either placebo or hormone will be initiated and continued for 135 minutes.

After 30 minutes of hormone infusion, a separate infusion of insulin (1.5mU/kg/min) will be initiated and continued for 60 minutes. Based on frequent bed-side plasma glucose measurements and an adjustable 20% glucose infusion, plasma glucose will be clamped at 2.5 mmol/l until the insulin infusion is terminated. Following this is a 45 minute recovery period, during which a minimum of glucose is infused, to ensure a steady rise from 2.5mmol/l to 3.5mmol/l.

After the study day, patients will receive a meal to prevent subsequent hypoglycemia.

The effects of each infusion will be evaluated with regards to glucagonotropic potency, as well as a series of exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Body mass index between 18-27kg/m2
* Type 1 diabetes (T1D) (diagnosed according to the criteria of the World Health Organization) with HbA1c<69 mmol/mol (<8.5%)
* T1D duration of 2-30 years
* C-peptide negative (stimulated C-peptide ≤ 100 pmol/l)
* Treatment with a stable basal-bolus or insulin pump regimen for ≥3 months
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Liver disease (ALAT and/or ASAT >2 times normal values) or history of hepatobiliary disorder
* Late microvascular complications except mild nonproliferative retinopathy
* Allergy or intolerance to ingredients included in the standardized meals
* Prior myocardial infarction or other cardiac events
* Any physical or psychological condition that the investigator feels would interfere with trial participation
* Treatment with any glucose-lowering drugs beside insulin

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Total glucagon response | 0-135minutes
  Difference in baseline subtracted area under the curve (bsAUC) for glucagon between study days with GIP[1-42], GIP[1-30] and placebo, respectively

SECONDARY OUTCOMES:
Glucagon response during insulin infusion | 30-90minutes
  Difference in bsAUC for glucagon between study days with GIP[1-42], GIP[1-30] and placebo, respectively during the insulin infusion
Glucagon response after blood glucose (BG) falls below 3.0 mmol/L | t[BG<3.0] and the following 30 minutes
  Difference in bsAUC for glucagon between study days with GIP[1-42], GIP[1-30] and placebo, respectively in the 30 minutes following a blood glucose of below 3.0 mmol/L
Glucagon response during recovery | 90-135minutes
  Difference in bsAUC for glucagon between study days with GIP[1-42], GIP[1-30] and placebo, respectively during the recovery period
Total insulin response | 0-135minutes
  Difference in plasma levels of insulin between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Total c-peptide response | 0-135minutes
  Difference in plasma levels of c-peptide between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Amount of glucose infused | 0-135minutes
  Difference in infusion rates for glucose between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in epinephrine | 0-135minutes
  Difference in plasma levels of epinephrine between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in norepinephrine | 0-135minutes
  Difference in plasma levels of norepinephrine between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in cortisol | 0-135minutes
  Difference in plasma levels of cortisol between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in growth hormone hormones | 0-135minutes
  Difference in plasma levels of growth hormone between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in Procollagen 1 Intact N-Terminal Propeptide (P1NP) | 0-135minutes
  Difference in plasma levels of P1NP between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in carboxy-terminal collagen crosslinks (CTX) | 0-135minutes
  Difference in plasma levels of CTX between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in blood pressure | 0-135minutes
  Difference in blood pressure between study days with GIP[1-42], GIP[1-30] and placebo, respectively
Difference in heart rate | 0-135minutes
  Difference in heart rate between study days with GIP[1-42], GIP[1-30] and placebo, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All published data will be made available to other researchers upon reasonable request